CLINICAL TRIAL: NCT00349960
Title: Once-Weekly Versus Once-Fortnightly Subcutaneous Epoetin Beta Administration in the Maintenance Phase of Anaemia Treatment in Haemodialyzed Patients
Brief Title: Epoetin Dosing Regimens in Haemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Romanian Society of Nephrology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3025
Record Dates: First submitted 2006-07-06; First posted 2006-07-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-02

CONDITIONS: Hemodialyzed Patients; Epoetin Treatment
Keywords: Erythropoiesis stimulating agent; Dosing frequency; Hemodialysis; Therapeutic equivalence

INTERVENTIONS:
Drug: NeoRecormon SC once-weekly versus once-every-other-week

SUMMARY:
Currently, less frequent than once weekly subcutaneous epoetin administration regimens were shown to be equally effective and safe as the once-weekly schedules in stable pre-dialyzed and peritoneal dialyzed patients Bioequivalence of once-every-two-weeks and once-weekly subcutaneous administration of the same total dose of epoetin beta for the maintenance phase of anemia treatment in stable, iron-replete, chronic hemodialyzed patients was therefore prospectively investigated.

two treatment schedules will be considered equivalent if the primary efficacy parameters will be simultaneously similar for both groups and in the predefined range of variation. Confidence intervals (CIs) will be used to compare groups. Since the target Hb in dialyzed patients is defined as 11g/dL (110 g/L) by the European Guidelines and as >10 g/dL (100 g/L) by the National Guidelines, with a recommended upper limit of 13 g/dL (130 g/L), the efficacy range for Hb in this study was predefined as 10-12 g/dL (100-120 g/L). The two treatment schedules will be considered to have similar efficacy if the mean Hb in Group 2w will not differ by more than ±0.5 g/dL (±5 g/L) compared to Group 1w during the assessment period. Once similar efficacy established, drug requirements will be compared calculating the ratio of the mean weekly epoetin doses in Group 2w/Group 1w. A range of 0.8 to 1.25 for the ratio is considered sufficient to define bioequivalence. Equivalence of drug usage in the two arms will be accepted if the whole 95% CI for this ratio will be within the above limits.

Lack of difference between group means does not imply similar distribution of treatment effects within each group. The individual hemoglobin change will be used to assess if response to treatment was similarly variable in the two arms. The change in Hb will be calculated for each patient as the difference between the mean Hb during the assessment period and the mean Hb during the baseline phase.

DETAILED DESCRIPTION:
Current European Best Practice Guidelines and the KDOQI Committee in the USA recommend preferential subcutaneous (SC) twice- to thrice-weekly epoetin administration. SC route significantly reduces epoetin requirements and therefore costs, compared to the intravenous (IV) route. Additionally, there is solid evidence showed once-weekly SC administration of epoetin beta to be equally efficient and well tolerated in hemodialyzed (HD) patients. Clinical studies suggest that the effects of epoetin alpha are sustained for more than one week, enabling less frequent schedules in pre-dialysis chronic kidney disease (CKD) patients. A recent European multicenter study in peritoneal dialysis (PD) patients confirmed that once-every-two-weeks SC epoetin beta is efficient and safe in the maintenance phase of anemia treatment for PD patients11. Thus, the optimum epoetin dosing regimen is still yet to be determined despite over a decade of clinical use.

All these data also suggest that the pharmacodynamic effects of epoetins could last longer than their plasma half-lives. The survival half-life of erythrocytes produced after exogenous epoetin administration is longer than that of erythrocytes produced in the absence of exogenous stimulation.

Apart of the academic interest, this issue has also direct implications on cost savings and increased patients' convenience. Furthermore, less frequent administration would reduce epidemiological hazards associated with populations at high risk of blood-borne viral infections such as hepatitis, particularly important in less developed countries, with a high prevalence of viral hepatitis infections (hepatitis B/C markers prevalences: 15.7%/45% in Romania versus 3%/13.5% in EuroDOPPS patients). While the potential benefits of less frequent dosing are clear, the efficacy and safety of such regimens must be fully investigated before adoption as standard treatment.

The present study investigates for the first time the equivalence of once-weekly versus once-every-two-weeks SC epoetin beta dosing regimens, in the maintenance phase of anemia therapy, in stable HD patients. The aim of the study is to assess whether once-every-other-week SC administration of the same total epoetin beta dose is as effective and as safe as SC once-weekly dosing.

In order to avoid a carry-over effect of the weekly schedule of epoetin treatment received prior to randomization, we defined a run-in period (weeks 1-12). Statistical analyses will be performed for the efficacy parameters determined during the assessment period only. The average for weeks 13-24 will be obtained by adding all values and dividing the sum by the number of time points for each patient during this period.

The two treatment schedules will be considered equivalent if the primary efficacy parameters will be simultaneously similar for both groups and in the predefined range of variation. Confidence intervals (CIs) will be used to compare groups. Since the target Hb in dialyzed patients is defined as 11g/dL (110 g/L) by the European Guidelines and as >10 g/dL (100 g/L) by the National Guidelines, with a recommended upper limit of 13 g/dL (130 g/L), the efficacy range for Hb in this study was predefined as 10-12 g/dL (100-120 g/L). The two treatment schedules will be considered to have similar efficacy if the mean Hb in Group 2w will not differ by more than ±0.5 g/dL (±5 g/L) compared to Group 1w during the assessment period. Once similar efficacy established, drug requirements will be compared calculating the ratio of the mean weekly epoetin doses in Group 2w/Group 1w. A range of 0.8 to 1.25 for the ratio is considered sufficient to define bioequivalence. Equivalence of drug usage in the two arms will be accepted if the whole 95% CI for this ratio will be within the above limits.

Lack of difference between group means does not imply similar distribution of treatment effects within each group. The individual hemoglobin change will be used to assess if response to treatment was similarly variable in the two arms. The change in Hb will be calculated for each patient as the difference between the mean Hb during the assessment period and the mean Hb during the baseline phase. The percentages of patients with target Hb and not requiring any increase in epoetin dose during the assessment period will be compared with chi-squared statistic.

The study is designed to detect a difference in Hb between the study groups of at least 0.5 g/dL (5 g/L), with a probability of 95% and a power of 0.9021, assuming a standard deviation of Hb in the HD population of 1.0 g/dL (10 g/L). A sample size of 85 patients is required in each arm of the trial. Since the study design includes epoetin doses variations in order to maintain target hemoglobin, it would have been expected that Hb would be constant and epoetin dose would vary. Therefore, the power calculations using epoetin doses as the outcome measure seem to be more appropriate. Considering a standard deviation of 39 IU/kg per week, a probability of 95% and a power of 90%, a sample size of 70 patients in each arm is required to detect a ± 20% difference in epoetin dose between groups. Because of an anticipated drop-out proportion of 15%, a minimum of 100 patients have to be enrolled in each group to satisfy both Hb and epoetin doses power conditions.

ELIGIBILITY:
Inclusion Criteria:

* adult age (≥18 years)
* at least 6 months on HD
* efficient HD (urea-equilibrated Kt/V >1.2, Daugirdas II equation)
* haemoglobin (Hb) levels above the Romanian recommended target of 10g/dL and stable (difference between the maximum and minimum values at three subsequent determinations ≤1.5g/dL)
* treatment with once-weekly SC epoetin beta for at least 2 months prior to enrollment
* serum ferritin level 80-800 ng/mL
* transferrin saturation 20-50%

Exclusion Criteria:

* poor blood pressure control (BP ≥140/90mmHg in spite of antihypertensive medication and fluid control by dialysis)
* cardiac failure or hepatic diseases (as defined by abnormal ALT and AST levels) or association of psychical disorders or other disturbances making the enrollment unacceptable, as judged by the physician
* hyperkalemia
* malnutrition (Subjective Global Assessment score B or C and/or serum albumin <4g/dL)
* acute infection or HIV infection
* significant inflammation (CRP >12 mg/L)
* severe hyperparathyroidism (iPTH >800 ng/mL)
* history of gastrointestinal bleeding
* > 5% variation in dry body weight in the last 6 months
* previously diagnosed folic acid and/or vitamin B12 deficiency
* neoplastic diseases
* other known causes of anaemia
* known hypersensibility to one of the administered drugs
* epilepsy
* pregnancy or lactation
* anti-viral treatment during the month preceding the inclusion
* immunosuppressive treatment or use of other medication known to influence erythropoiesis 4 weeks before the enrollment
* participation in another clinical trial 4 weeks prior to enrollment
* need for blood transfusions within 8 weeks prior to enrollment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-03; Study Completion 2005-12

PRIMARY OUTCOMES:
hemoglobin level in the assessment period (average of all values from weeks 13-24)
weekly epoetin beta dose per dry body weight in the assessment period (average of all values from weeks 13-24)

SECONDARY OUTCOMES:
the percentage of patients maintaining target Hb without any increase in epoetin dose during the assessment period;
the difference between the average Hb levels during the assessment period versus the baseline phase;
the difference between the average weekly epoetin beta dose during the assessment period versus the baseline phase.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Mircescu Mircescu, Professor, Study Director — Romanian Society of Nephrology
Locations (9):
- Romania (9):
  - "Dr Carol Davila" Teaching Hospital of Nephrology, Bucharest
  - "Sf. Ioan Nou" Clinical Hospital, Nephrology and Dialysis Department, Bucharest
  - Dialysis Centre, "Fundeni" Clinical Institute, Bucharest, Bucharest
  - Dialysis Centre, Army Medical Diagnosis and Treatment Centre, Bucharest
  - Nephrology and Dialysis Clinic, Cluj Clinical County Hospital, Cluj-Napoca
  - Nephrology and Dialysis Clinic, Craiova Clinical County Hospital, Craiova
  - Dialysis and Transplantation Center, "CI Parhon" University Hospital, Iași
  - Nephrology and Dialysis Department, Dâmboviţa County Hospital, Târgovişte
  - Dialysis and Renal Transplantation Centre, Timisoara County Hospital, Timișoara